CLINICAL TRIAL: NCT06763419
Title: Internal Photobiomodulation For Management Of Temporomandibular Joint Internal Derangement: A Randomized Clinical Trial
Brief Title: Internal Photobiomodulation For Management Of Temporomandibular Joint Internal Derangement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0828-12/2023
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External low level laser therapy (Experimental)
  Interventions: Device: External low level laser therapy
- Internal low level laser therapy (Active Comparator)
  Interventions: Device: Internal low level laser therapy

INTERVENTIONS:
Device: External low level laser therapy — Patients received 8 sessions of external diode laser (635 nm).
  Arms: External low level laser therapy
Device: Internal low level laser therapy — Patients received 8 diode laser (635 nm) sessions applied internally
  Arms: Internal low level laser therapy

SUMMARY:
Aim of the study was to compare the efficacy of internal versus external photobiomodulation (PBM) in the management of patients with TMJ internal derangements (TMJ-ID).

ELIGIBILITY:
Inclusion Criteria:

* Painful click at temporomandibular joint (TMJ) area.
* Pain at the lateral pterygoid muscle.
* Presence of full or nearly full complement of natural teeth with acceptable occlusion

Exclusion Criteria:

* Patients who have radiographic evidence of degenerative conditions of TMJ.
* Patients under current dental or physical therapy that could affect TMD.
* History of recent trauma.
* The presence of systemic diseases (i.e. rheumatoid arthritis, osteoarthritis).
* Pregnant and lactating females.
* Presence of open bite.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain level assessment using Visual Analogue Scale | after one month from the last laser session
  All patients will be evaluated subjectively through Visual Analogue Scale (VAS) to clinically assess the pain intensity with ratings between 0 for pain-free and 10 for maximum pain
Oral health-related quality of life using OHIP-TMD | after one month from the last laser session
  Oral health-related quality of life will be assessed using OHIP-TMD, a 22-item temporomandibular disorder-specific version of the Oral Health Impact Profile (OHIP).
  Each item in the OHIP-TMDs is scored on a Likert scale, often ranging from: 0 (Never) to 4 (Very often). For each respondent, the scores for all 22 items are summed to create a total score. The total score ranges from 0 to 88, where higher scores indicate a greater negative impact on oral health-related quality of life.
Maximum mouth opening evaluation using the Miller index | after one month from the last laser session
  The Miller Index is calculated as a ratio of the observed maximum interincisal distance (distance between the edges of the upper and lower incisors when the mouth is fully open) to the patient's height. This provides a normalized measure of mouth opening relative to body stature.
  Miller Index= Maximum Interincisal Distance (mm)/Height (cm)
  Normal Range: A typical Miller Index is around 1.6 to 1.7 mm/cm in healthy individuals. This means that for every centimeter of height, the expected mouth opening is about 1.6 to 1.7 mm.
  Deviations:
  * Lower than Normal: May indicate restricted mouth opening (e.g., trismus, TMDs, fibrosis, ankylosis).
  * Higher than Normal: May occur in conditions involving hypermobility.

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen Rady, PhD, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Mariam M Bahgat, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Aly Atteya, PhD, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Hoda MA Abdel-Naby, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt